CLINICAL TRIAL: NCT04363541
Title: A Multicenter, Open-label, Parallel-group, Randomized, Adaptive Trial to Evaluate Local Thermotherapy in Patients With Mild-to-moderate COVID-19, to Prevent Disease Progression
Brief Title: Local Thermotherapy for Patients With Mild-to-moderate COVID-19
Acronym: TherMoCoV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Perinatologia (Other Government)
Collaborators: Direccion General de Calidad y Educacion en Salud (Unknown); Instituto Mexicano del Seguro Social (Other Government); Hospital Regional de Alta Especialidad Juan Graham Tabasco (Unknown); Hospital Dr. Ángel Leaño (Unknown); National Polytechnic Institute, Mexico (Other); Universidad Juárez Autónoma de Tabasco (Other)
Responsible Party: Principal Investigator, Norma del Carmen Galindo-Sevilla, Principal Investigator, Instituto Nacional de Perinatologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1250-7416
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: COVID-19; Thermotherapy
Keywords: SARS-CoV-2; Hyperthermia
MeSH Terms: conditions — COVID-19; Hyperthermia

STUDY DESIGN:
Intervention Model Description: The application of an electric chest pad. The use of an electric cushion was chosen because it is designed to be used in human thermal therapy. The electric cushion provides continuous 90 minutes of regulated heat, with enough penetration to raise the external temperature of the area to 40-42 ° C.
  It is a therapy designed to detain disease progression. It is not expected to have an effect on concomitant microorganisms such as bacteria or opportunists such as Candida albicans, so that when the concomitant infection is suspected, the antibiotic of choice should be given or continued, depending on the nature of the infection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Thermotherapy (Experimental): Electric heat pad applied in the thorax for 90 minutes, twice daily, for 5 days.
  + Usual in-hospital care
  Interventions: Device: Electric pad for human external pain therapy
- Control (No Intervention): Usual in-hospital care

INTERVENTIONS:
Device: Electric pad for human external pain therapy — An electric pad for local heat production will be put on the back of the patient for two hours
  Arms: Thermotherapy

SUMMARY:
The etiological agent of the current pandemic is a (+)ssRNA virus. SARS-CoV-2 is infecting thousands of people in the world with a fatality rate that varies from 0.1 to 5% in affected countries, thereby causing enormous economic losses. Few antibiotics have shown any efficacy in their combat, but have not yet proven adequate to stop the spread of the disease, nor are there any approved vaccines at the moment. From experiments in plants ongoing infections by RNA viruses, using thermotherapy, which is the application of heat at a temperature between 35-43 °C, the investigators know that raising the temperature affects the transcription of viral proteins due to the formation of small RNA molecules that interrupt the replication process by grouping in specific regions of the RNA molecule, preventing and inhibiting transcription. These small molecules are called small interfering RNAs (siRNAs). This feature has been used through thermotherapy in humans to combat the rapid replication of cells (i.e. cancer cells), attack cells infected by RNA viruses, and in the treatment of some parasitic infections.There are various commercially available devices for thermotherapy use in humans; they are mainly being used to ease muscle pain. They work by increasing the temperature in the range recommended for thermotherapy in humans 39-43 ° C. Therefore, the investigators consider this treatment modality can be used to aid in the elimination of SARS-CoV-2 from the human body, decreasing viral load, which could allow the immune system time for its control and elimination.

DETAILED DESCRIPTION:
Considering the nature of the causative agent of COVID-19, a (+)ssRNA virus, the investigators propose the use of thermotherapy as a modality for viral containment, thereby preventing the progression of the infection to severe cases. The investigators consider applying the intervention with thermotherapy mainly as an adjuvant therapy in high-risk patients. The most accessible thermotherapy delivery method the investigators have identified is the use of an electric chest pad for its wide and known clinical use, including its recommended use for patients with arthritis. The intensity of temperature delivered by the electric cushion should be placed on the first level (lowest level), to avoid discomfort to the patient. The electric cushion provides a continuous hour of regulated heat, with enough penetration to raise the external temperature of the area to 40-42 ° C, a temperature range at which facilitation of elimination of the virus is expected.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with symptoms of COVID-19 (fever, headache, cough, sore throat, myalgias, arthralgias, shortness of breath, anosmia, fatigue, diarrhea, vomit, or conjunctivitis) meeting criteria for mild or moderate COVID-19 according to the following criteria:

   1. Mild COVID-19: With or without mild pneumonia. Peripheral oxygen arterial saturation (SaO2) greater than or equal to 94% (90% in Mexico City and Guadalajara) at room air. Does not meet criteria of moderate, severe, or critical COVID-19.
   2. Moderate COVID-19: Patient with pneumonia and risk factors for disease progression; meeting all the following: Shortness of breath, peripheral oxygen arterial saturation (SaO2) greater than or equal to 94% (90% in Mexico City and Guadalajara) with a maximum 3 L/min of supplementary oxygen, does not meet criteria for severe, or critical COVID-19.
2. Patient with less than or equal to 5 days from symptom onset
3. Participant understands the intervention and procedures and accepts randomization.

Exclusion Criteria:

1. Suspected or confirmed pregnancy at evaluation
2. Severe decompensation of any of the patient's underlying diseases
3. Previous diagnosis of COVID-19 with complete resolution of symptoms for at least 2 days.
4. Patients meeting criteria for severe or critical COVID-19 at evaluation:

   1. Severe COVID-19 - Patient with ≥1 of the following: tachypnea (≥30 breaths per minute), peripheral oxygen arterial saturation (SaO2) less than or equal to 93% (89% in Mexico City and Guadalajara) with a maximum 3 L/min of supplementary oxygen (patients requiring ≥4 L/min will be considered to have progressed to severe COVID-19), or PaO2/FiO2 ratio <300.
   2. Critical COVID-19 - Patient with ARDS, shock, multiorgan failure, or any other condition requiring admission to an intensive care unit.

Elimination Criteria:

1. Participant retires consent to participate in the study
2. Patient requiring ≥4 L/min of supplementary oxygen in the 24 hours of hospitalization (in the case that randomization occurred in the first 24 hours of hospitalization)
3. Two negative tests against SARS-CoV-2 (a sequential diagnostic strategy will be implemented to reduce losses due to false negative tests).
4. Patient that do not tolerate thermotherapy and requests to stop receiving the intervention.
5. Transfer to another medical unit in the first 5 days of inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Progression of disease (composite outcome) | 28 days
  Progression to any of the following:
  1. Severe COVID-19 - Patient with ≥1 of the following: tachypnea (≥30 breaths per minute), peripheral oxygen arterial saturation (SaO2) less than or equal to 93% (89% in Mexico City and Guadalajara) with a maximum 3 L/min of supplementary oxygen (patients requiring ≥4 L/min will be considered to have progressed to severe COVID-19), or PaO2/FiO2 ratio <300.
  2. Critical COVID-19 - Patient with ARDS, shock, multiorgan failure, or any other condition requiring admission to an intensive care unit.
  3. Death

SECONDARY OUTCOMES:
Mortality at day 15 | 15 days
  Proportion of participants deceased by day 15 after enrollment
Mortality at day 28 | 28 days
  Proportion of participants deceased by day 28 after enrollment
Time to progression to severe COVID-19 | Up to 33 days
  Days from symptom onset to progression to severe COVID-19
Time to progression to critical COVID-19 | Up to 33 days
  Days from symptom onset to progression to critical COVID-19
Hospitalization time | Up to 33 days
  In-hospital stay in days
Percentage of participants at each clinical status in the Ordinal Scale at Day 15 | 15 days
  Ordinal scale of 7 categories: 1) Not hospitalized, without limitations on daily activities; 2) Not hospitalized, with limitations on daily activities; 3) Hospitalized, not requiring supplementary oxygen; 4) Hospitalized, requiring low-flow supplementary oxygen; 5) Hospitalized, requiring supplementary oxygen with high-flow nasal cannula or non-invasive ventilation; 6) Hospitalized, under invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 7) Death
Percentage of participants at each clinical status in the Ordinal Scale at Day 28 | 28 days
  Ordinal scale of 7 categories: 1) Not hospitalized, without limitations on daily activities; 2) Not hospitalized, with limitations on daily activities; 3) Hospitalized, not requiring supplementary oxygen; 4) Hospitalized, requiring low-flow supplementary oxygen; 5) Hospitalized, requiring supplementary oxygen with high-flow nasal cannula or non-invasive ventilation; 6) Hospitalized, under invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 7) Death
Time (days) to last requiring supplementary oxygen according to modality | 28 days
  Modalities: 1) Simple nasal cannula or face mask; 2) Face mask with reservoir; 3) High-flow nasal cannula; 4) Non-invasive mechanical ventilation; 5) Invasive mechanical ventilation
Change in National Early Warning Score 2 (NEWS-2) with respect to baseline | Days 1, 5, 15, and 28
  Change in the National Early Warning Score 2 (NEWS-2) with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.
  This score evaluates 7 parameters (respiratory rate, peripheral arterial oxygen saturation, supplementary oxygen requirements, systolic arterial blood pressure, heart rate, consciousness, and body temperature). Assigned values for every parameter may range from 0 to 3 points, except for supplementary oxygen for which possible values are 0 (not requiring supplementary oxygen) and 2 (requiring supplementary oxygen). The total sum of points for this score may range from 0 to 20 points. Higher scores reflect increasing clinical deterioration.
Proportion of patients requiring invasive mechanical ventilation | 28 days
  Proportion of patients requiring invasive mechanical ventilation during the entire follow-up period
Proportion of patients requiring admission to intensive care unit (ICU) | 28 days
  Proportion of patients requiring admission to intensive care unit (ICU) during the entire follow-up period
Time to requiring invasive mechanical ventilation | Up to 33 days
  Days from symptom onset to progression to requiring invasive mechanical ventilation
Time to requiring admission to intensive care unit (ICU) | Up to 33 days
  Days from symptom onset to requiring admission to intensive care unit (ICU)
Proportion of patients with adverse events according to outcome | 28 days
  * Severe: Causes death of the patient, puts the patient's life at risk in the moment of occurrence, requires hospitalization or prolongs hospitalization, causes persistent or significant disability.
  * Non-severe adverse events: Do not meet the previously outlined criteria.
Proportion of patients with adverse events according to severity | 28 days
  * Mild (Grade 1): Present with easily tolerated signs and symptoms, do not need specific treatment, do not prolong hospitalization, nor require suspension of the intervention
  * Moderate (Grade 2): Interfere with daily activities (school or work), do not directly threaten life, require specific pharmacological treatment, and do not necessarily require suspension of the intervention.
  * Severe (Grades 3, 4, and 5): Interfere with daily activities (school and work), require pharmacological treatment and suspension of the intervention.
Proportion of patients with adverse events according to causality | 28 days
  * Certain
  * Probable
  * Possible
  * Uncertain
  * Unclassifiable
Proportion of patients tolerating the intervention (no comparison) | 5 days
  Proportion of patients tolerating the intervention (number of sessions and minutes per session).

OTHER OUTCOMES:
Comparison of laboratory parameters with respect to baseline (units: 10^3/microliter) | Days 1, 5, 15, and 28
  Change in laboratory parameters with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.
  Parameters to be included are: total leucocytes, neutrophils, lymphocytes, monocytes, and platelets
Comparison of laboratory parameters with respect to baseline (units: milligrams/deciliter) | Days 1, 5, 15, and 28
  Change in laboratory parameters with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.
  Parameters to be included are: glucose, urea, blood urea nitrogen, creatinine, total bilirubin, direct bilirubin, and indirect bilirubin.
Comparison of laboratory parameters with respect to baseline (units: grams/deciliter) | Days 1, 5, 15, and 28
  Change in laboratory parameters with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.
  Parameters to be included are: hemoglobin, and albumin
Comparison of laboratory parameters with respect to baseline (units: milligrams/liter) | Days 1, 5, 15, and 28
  Change in laboratory parameters with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.
  Parameters to be included are: C-reactive protein
Comparison of laboratory parameters with respect to baseline (units: nanograms/milliliter) | Days 1, 5, 15, and 28
  Change in laboratory parameters with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.
  Parameters to be included are: D-dimer, and procalcitonin
Comparison of laboratory parameters with respect to baseline (units: International Units/liter) | Days 1, 5, 15, and 28
  Change in laboratory parameters with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.
  Parameters to be included are: aspartate aminotransferase (AST), alanine aminotransferase (ALT), lactate dehydrogenase (LDH), and creatinine phosphokinase (CPK).
Comparison of laboratory parameters with respect to baseline (ratio: no units) | Days 1, 5, 15, and 28
  Change in laboratory parameters with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.
  Parameters to be included are: neutrophil-to-lymphocyte ratio, and international normalized ratio (INR).
Comparison of laboratory parameters with respect to baseline (units: percent) | Days 1, 5, 15, and 28
  Change in laboratory parameters with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.
  Parameters to be included are: hematocrit
Comparison of laboratory parameters with respect to baseline (units: seconds) | Days 1, 5, 15, and 28
  Change in laboratory parameters with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.
  Parameters to be included are: prothrombin time (PT), and partial thromboplastin time (PTT)
Comparison of laboratory parameters with respect to baseline (units: millimeters/hour) | Days 1, 5, 15, and 28
  Change in laboratory parameters with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.
  Parameters to be included are: erythrocyte sedimentation rate (ESR)
Comparison of cytokine levels with respect to baseline | Days 1, 5, 15, and 28
  Change in cytokine levels with respect to baseline (Day 1), measured at day 5 for all patients, and days 15 & 28 only for patients that remain hospitalized.

CONTACTS AND LOCATIONS:
Overall Officials: Norma del Carmen Galindo Sevilla, PhD, Principal Investigator — Instituto Nacional de Perinatología; Javier Mancilla-Galindo, MBBS, Study Director — Instituto Nacional de Cardiología
Locations (3):
- Mexico (3):
  - Hospital Dr. Ángel Leaño, Guadalajara, Jalisco
  - Hospital Regional de Alta Especialidad "Dr. Juan Graham Casasus", Villahermosa, Tabasco
  - Unidad Temporal Movil COVID-19 Autódromo Hermanos Rodríguez IMSS, Mexico City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu J, Zhang X, Zhang F, Hong N, Wang G, Wang A, Wang L. Identification and characterization of microRNAs from in vitro-grown pear shoots infected with Apple stem grooving virus in response to high temperature using small RNA sequencing. BMC Genomics. 2015 Nov 16;16:945. doi: 10.1186/s12864-015-2126-8. PMID 26573813
- [Background] Wang MR, Cui ZH, Li JW, Hao XY, Zhao L, Wang QC. In vitro thermotherapy-based methods for plant virus eradication. Plant Methods. 2018 Oct 6;14:87. doi: 10.1186/s13007-018-0355-y. eCollection 2018. PMID 30323856
- [Background] Zhu LL, Gao XH, Qi R, Hong Y, Li X, Wang X, McHepange UO, Zhang L, Wei H, Chen HD. Local hyperthermia could induce antiviral activity by endogenous interferon-dependent pathway in condyloma acuminata. Antiviral Res. 2010 Nov;88(2):187-92. doi: 10.1016/j.antiviral.2010.08.012. Epub 2010 Aug 24. PMID 20797409
- [Derived] Mancilla-Galindo J, Kammar-Garcia A, Mendoza-Gertrudis ML, Garcia Acosta JM, Nava Serrano YS, Santiago O, Torres Vasquez MB, Martinez Martinez D, Fernandez-Urrutia LA, Robledo Pascual JC, Narvaez Morales ID, Velasco-Medina AA, Mancilla-Ramirez J, Figueroa-Damian R, Galindo-Sevilla N. Regional moderate hyperthermia for mild-to-moderate COVID-19 (TherMoCoV study): a randomized controlled trial. Front Med (Lausanne). 2023 Dec 22;10:1256197. doi: 10.3389/fmed.2023.1256197. eCollection 2023. PMID 38188344